CLINICAL TRIAL: NCT00458614
Title: Lansoprazole Disposition in Young Children With Cystic Fibrosis
Brief Title: Pharmacokinetic Study of Lansoprazole in Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPRU-10840
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole

SUMMARY:
The disposition of a number of drugs has been reported to be altered in patients with Cystic Fibrosis (CF). Changes in pharmacokinetic parameters observed included increased volumes of distribution and increased clearance of renally eliminated drugs. The purpose of this this study is to characterize the pharmacokinetics of IV lansoprazole and its metabolites in normal healthy children and children with Cystic Fibrosis (CF) ages 2 to < 10 years. It is suspected that children with CF will have a more rapid clearance as compared to healthy children.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) impacts 1:2500 Caucasian newborns and results from a defect in the cystic fibrosis transmembrane conductance regulator chloride channel (CFTR) responsible for electrolyte regulation. Between 25 to 81% of the CF population have gastro-esophageal reflux disease (GERD), and proton pump inhibitors (PPIs) are frequently prescribed for this condition. Moreover, PPIs are commonly used in patients with CF to allow for better gastric acid stabilization so that pancreatic enzyme efficacy is optimized and nutritional status is improved. Lansoprazole is a PPI that is widely used for acid-related disorders including GERD.

The disposition of a number of drugs has been reported to be altered in CF. Changes in pharmacokinetic parameters observed in patients with CF include increased volumes of distribution and increased clearance of renally eliminated drugs. To date, the pharmacokinetics of PPIs in patients with CF have not been characterized.

This study is a pilot study to evaluate and compare the pharmacokinetics of a single dose of IV lansoprazole in CF and normal children 2 to < 10 years of age. A goal of 12 evaluable subjects ranging from 2 to < 10 years of age including both males and females with CF ∆F508 genotype will be recruited from CF clinic or inpatient. As a comparison group, six evaluable subjects who are normal, healthy children of similar demographic profile (age, gender, and race) will be recruited.

After informed consent/assent is obtained, screening procedures will be completed within 30 days of study participation. The pre-study screen includes an age-appropriate physical exam, medical history (current medication/herbal use), vital signs (non-crying sitting blood pressure and heart rate), height, weight, AST, ALT, and CBC. Subjects will be studied during a current hospitalization or scheduled for an approximately 12-hour study visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have the diagnosis of CF with the ∆F508 genotype (hetero- or homozygous) or who are normal and healthy as determined by the principal investigator, have in the past year received a H2 receptor antagonist, PPI, or antacid, and do not meet any of the exclusion criteria.
* Subjects of either gender and all races and ethnicity age 2 to < 10 years.
* Written informed consent from parent or guardian who has sufficient intellectual capacity to understand the study and adhere to the procedures and as applicable (i.e., subjects ≥ 7 years of age), subject assent.

Exclusion Criteria:

* Refusal of informed consent/assent by the parent/caregiver and child > 7 years of age.
* Body weight less than 10 kg.
* Three or more hospitalizations during the preceding year.
* Severe liver dysfunction (AST & ALT > 3 times the upper normal limit).
* Clinically significant (determined by investigator) alterations in hemoglobin and/or hematocrit.
* Pregnancy or lactation.
* Concurrent therapy with agents other than a PPI that are known to be CYP2C19 substrates within 2 weeks of study drug administration
* PPI use within 48 hours of study drug administration.
* Acute change in health status within 72 hours of study drug administration.
* Allergy or hypersensitivity to lansoprazole or to other proton pump inhibitors

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18
Dates: Start 2006-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Examine the PK enantiomers of IV lansoprazole and metabolites, in normal children and children with CF.

SECONDARY OUTCOMES:
To compare the differences in the PK enantiomers of IV lansoprazole and metabolites, between children with CF and normal healthy children
Examine the PK enantiomers of IV lansoprazole and metabolites in relationship to CYP2C19 genotype in children with CF and normal healthy children
To assess the effects of ontogeny on IV lansoprazole drug disposition

CONTACTS AND LOCATIONS:
Overall Officials: Holly D Maples, Pharm.D., Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital Little Rock, Little Rock, Arkansas, United States